CLINICAL TRIAL: NCT06192225
Title: Peri-operative Slow-paced Breathing - a Non-invasive Technique to Reduce Anxiety in Breast Cancer Surgery Patients
Brief Title: Peri-operative Slow-paced Breathing to Reduce Anxiety in Breast Cancer Surgery Patients
Acronym: SlowPACE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N23SLO
Record Dates: First submitted 2023-06-22; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-10

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single center, two-group, prospective, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slow PACE arm (Experimental): The intervention consists of performance of pre-trained guided Slow PACE breathing by the patient at induction of anesthesia for breast cancer surgery.
  Interventions: Behavioral: pre-trained guided slow paced breathing (~6 breaths per minute)
- Control arm (No Intervention): Care as usual

INTERVENTIONS:
Behavioral: pre-trained guided slow paced breathing (~6 breaths per minute) — Slow PACE breathing
  Arms: Slow PACE arm

SUMMARY:
The purpose of this single-center trial is to examine the effects of a slow-breathing technique performed at induction of anesthesia in patients undergoing surgery for breast cancer on anxiety, scored by Spielberger's State-Trait Anxiety Inventory, state scale (STAI-S),13 compared to usual care.

DETAILED DESCRIPTION:
Rationale: In the perioperative period anxiety for anesthesia and the surgical procedure is common. Breast cancer surgery patients have a higher level of anxiety compared to other patients undergoing (cancer) surgery. Relaxation techniques, like breath focus with deep belly breathing are easy to learn and can have a beneficial effect on postoperative anxiety, pain, and postoperative nausea and vomiting (PONV), but the quality of evidence is low. Slow paced breathing at a frequency of 6 breaths per minute can possibly increase vagal activation, decrease anxiety, reduce mean blood pressure, and postoperative pain.

The investigators aim to apply a pre-trained slow paced breathing technique at induction of anesthesia for surgery, to reduce perioperative anxiety and to explore effects on pre-operative blood pressure, per-operative need of hypnotics, postoperative pain and opioid use, PONV and patient satisfaction.

Objective: This study aims to examine the effects of guided slow paced breathing performed at induction of anesthesia in patients undergoing surgery for breast cancer on anxiety, scored by Spielberger's State-Trait Anxiety Inventory, State scale (STAI-S), compared to usual care.

Study design: Single center, two-group, prospective, randomized controlled trial Study population: patients scheduled for surgery for breast cancer in the Antoni van Leeuwenhoek Hospital.

Intervention: Performance of pre-trained guided slow paced breathing by the patient at induction of anesthesia for breast surgery.

Main study parameters: Anxiety scored by Spielberger's State Anxiety Inventory (STAI-S) Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There are no risks related to the intervention. Participants randomized in the intervention group are trained in slow paced breathing after inclusion and asked to practice the technique daily until the day of surgery. All participants are asked to complete three questionnaires at baseline, and two short questionnaires on the day of surgery and at day 1.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Undergoing surgery for breast cancer in the Antoni van Leeuwenhoekziekenhuis

Exclusion Criteria:

* Age < 18 years
* ASA ≥ 4
* History of severe pulmonary illness: severe asthma or severe chronic obstructive pulmonary disease (COPD) GOLD III or IV
* Known or suspected severe psychiatric disorder
* Unable to give written or oral informed consent
* Patient refusal
* Not able to understand Dutch
* No internet access
* Visual or hearing impairments interfering with reading and listening to the online material

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Population of patients with breast cancer
Enrollment: 150 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-02 (Estimated)

PRIMARY OUTCOMES:
Peri operative anxiety | 2 weeks
  The present study aims to examine the effects of pre-trained guided Slow PACE breathing performed at induction of anesthesia in patients undergoing surgery for breast cancer on anxiety, scored by Spielberger's State-Trait Anxiety Inventory, state scale (STAI-S), compared to usual care.
  The total score ranging from 20 to 80. Higher scores indicate higher levels of anxiety symptoms. A cut-off score of 40 is commonly used to define probable clinical levels of anxiety.

SECONDARY OUTCOMES:
mean blood pressure before induction | 10 minutes
  MAP (mmHg)
need of hypnotics during induction | 10 minutes
  total dose of hypnotics (propofol in milligrams)
post-operative pain | post-operative on recovery (1-2hours)
  visual analoge score (VAS) for pain, 0-10 points. A VAS score > 4 indicates the need of more pain medication
post-operative need of opioids | post-operative on recovery (1-2hours)
  Mean cumulative intravenous opioid dose administered during admission in the recovery room - converted to morphine equivalent dose (MEQ)
postoperative nausea and vomiting (PONV) | post-operative on recovery (1-2hours)
  Y/N
patient satisfaction | 5 minutes on postoperative day 1
  scale of 0 (extremely unsatisfied) to 10 (extremely satisfied)
Anxiety trait scored by Spielberger's State Anxiety Inventory (STAI-T)13 at baseline | once at baseline, duration 10 minutes
  4-point scale ranging from 1 (not at all) to 4 (very much so), with the total score ranging from 20 to 80. Higher scores indicate higher levels of anxiety symptoms. A cut-off score of 40 is commonly used to define probable clinical levels of anxiety. The STAI-T will give an estimation of patients at high risk for anxiety.
Hospital Anxiety and Depression Scale (HADS-A) | once at baseline, duration 10 minutes
  A questionnaire for detecting states of anxiety and depression in a hospital setting. The HADS-A is the anxiety subscale that consists of seven items. Each item is rated on a 4-point scale (ranging from 0 = no not at all, to 3 = yes definitely), for a total score ranging from 0 to 21. A subscale score above 8 denotes anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Antoni van Leeuwenhoek hospital, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No
currently there are no other researchers

REFERENCES:
- [Background] Spielberger, C.D. (2010). State-Trait Anxiety Inventory. In The Corsini Encyclopedia of Psychology (eds I.B. Weiner and W.E. Craighead).
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT06192225/Prot_SAP_000.pdf